CLINICAL TRIAL: NCT01932008
Title: Evaluation of the Bone Mineral Density and Muscle Mass in Patients Post Coronary Artery Bypass Graft Surgery With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH-IRB-100110-F
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Bypass Graft; Chronic Kidney Disease
Keywords: Coronary artery bypass grafting; Chronic kidney disease; Body composition; Physical activity; Physical function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purposes of this study are: (1) to compare the body composition, physical activity, physical function, and quality of life between patients with and without CKD after CABG; and (2) to analyze the relationships among body composition, physical activity, and physical function in this population. It is expected that patients after CABG with CKD have the worse body composition, physical function, and quality of life than patients after CABG without CKD; and patients with higher physical activity levels have the better body composition, physical function, and quality of life.

DETAILED DESCRIPTION:
It has been reported that cardiac disease and renal disease frequently coexisted. Recently, the term cardiorenal syndrome was used to describe the interaction between heart and kidney. Chronic kidney disease (CKD) has become increasingly recognized as an independent risk factor of cardiovascular disease, and the cardiovascular disease is one of most severe complication in patients with CKD. Previous studies have showed the changes in body composition, physical inactivity, decreased physical function, and poor quality of life existed in patients with either cardiovascular disease or CKD. Patients concomitant with cardiovascular disease and kidney insufficiency were expected to significantly increase physical dysfunction. However, few studies addressed on these alterations in patients after coronary artery bypass grafting (CABG) with CKD were reported.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing CABG without valve surgery
* chronic kidney disease(matched group: without CKD)

Exclusion Criteria:

1. heart transplantation or redo CABG
2. amputation,
3. cerebrovascular disease or any others disease with limbs dysfunction,
4. lung deficit,
5. cancer,
6. cognitive disorders.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent CABG at the Department of Cardiovascular Center at Far-Eastern Memorial Hospital since January 2000 were selected for recruitment to this study.Thirty male patients after CABG with CKD and 30 matched controls were recruited (ages between 40-75 years old).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
lean body mass and body fat | The participants were followed at one time points after operation in past 10 years
  All the subjects underwent dual-energy x-ray absorptiometry(DEXA) examination for body composition evaluation. The lean body mass and body fat were examined by DEXA.

SECONDARY OUTCOMES:
physical activity | The participants were followed at one time points after operation in past 10 years
  The level of physical activity was evaluated by the self-administrated long form of the International Physical Activity Questionnaire, which was permitted by the Bureau of Health Promotion, Department of Health, R.O.C.(Taiwan). It is an instrument that estimates the weekly time spent on the performance of physical activities according to intensity, in different contexts of life (workplace, household tasks, transport and leisure). Reported minutes per week in each category were weighted by a metabolic equivalent (MET; multiples of resting energy expenditure).
physical function | The participants were followed at one time points after operation in past 10 years
  The outcome measures of physical function included grip strength, 30-second chair stand test, and six-minute walk test(6MWT).
quality of life | The participants were followed at one time points after operation in past 10 years
  QOL was measured using abbreviated version of the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire. The original WHOQOL-BREF comprised 26 questions and included four domains: physical, psychological, social relationships, and environment. The WHOQOL-BREF scale has been adapted for Taiwan and added two questions appropriate for Taiwanese culture.